CLINICAL TRIAL: NCT06689644
Title: Effect of a Plant-based Nootropic Supplement on Perceptual Decision-making and Brain Network Interdependencies: a Randomised, Double-blinded and Placebo-controlled Study.
Brief Title: Effect of a Plant Based Nootropic on Perceptual Decision Making.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Dr Andrea Utley, Professor, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: AUtley
Record Dates: First submitted 2024-11-13; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Cognitive Enhancement
Keywords: Perceptual decision-making; Cognitive enhancement; Nootropics; EEG; Brain health
MeSH Terms: interventions — Nootropic Agents; Ginkgo Extract; Nicergoline; Piracetam; Electroencephalography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): This group will receive the nootropic supplement for 60 days.
  Interventions: Dietary Supplement: Nootropics (ginkgo biloba, nicergoline, piracetam, or others); Behavioral: Perceptual decision-making performance; Device: Electroencephalography
- Control group (Placebo Comparator): This group will receive a placebo supplement for 60 days
  Interventions: Dietary Supplement: Placebo; Behavioral: Perceptual decision-making performance; Device: Electroencephalography

INTERVENTIONS:
Dietary Supplement: Nootropics (ginkgo biloba, nicergoline, piracetam, or others) — Commercially available product: Mind lab pro
  Arms: Experimental group
Dietary Supplement: Placebo — A cellulose commonly used as a bulking agent in supplement products
  Arms: Control group
Behavioral: Perceptual decision-making performance — A computerised cognitive task involving rapid visual categorisation of images
Device: Electroencephalography — Brain signals are recorded from a 64 channel EEG system during the cognitive task

SUMMARY:
Nootropics are a group of medicinal substances purported to improve important cognitive functions such as learning, focus and memory. Many of these substances have demonstrated beneficial effects on cognitive performance and overall health. However, a thorough understanding of how these substances and their synergistic effects in the form of a supplement may benefit fundamental brain processes is currently lacking. In the current study, we will investigate the effects of a plant-based, nootropic supplement (https://uk.mindlabpro.com/) on perceptual decision-making (i.e. the ability to make rapid decisions based on sensory stimuli) in healthy adult participants.

DETAILED DESCRIPTION:
Participants will perform a computerised cognitive task assessing their perceptual decision-making pre- and post- 60 days of continuous supplementation with either a plant-based nootropic supplement (Mind Lab pro) or placebo. During testing, electroencephalography (EEG) signals will be captured simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility screening of participants was guided by the following inclusion criteria: (i) be between 20-59 years old, (ii) be right-handed and (iii) be able to cease taking other dietary supplements for two months.

Exclusion Criteria:

* Exclusion criteria included: (i) currently consuming a nootropic supplement, (ii) any known musculoskeletal, or neurological medical conditions or cognitive impairments (iii) have a known diagnosis of epilepsy/history of seizures and (iv) have a known hearing or visual condition that affects daily life function.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Perceptual decision-making performance | Pre- and post- 60 days of supplementation
  Choice accuracy and reaction times

SECONDARY OUTCOMES:
Brain network interdependencies | Pre- and post- 60 days of supplementation
  Patterns extracted from brain signals using electroencephalography

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Delis, Principal Investigator — University of Leeds
Locations (1):
- Faculty of Biological sciences, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No further investigations will take place using this data with anyone outside of the current research group

REFERENCES:
- [Derived] O'Reilly D, Bolam J, Delis I, Utley A. Effect of a Plant-Based Nootropic Supplement on Perceptual Decision-Making and Brain Network Interdependencies: A Randomised, Double-Blinded, and Placebo-Controlled Study. Brain Sci. 2025 Feb 21;15(3):226. doi: 10.3390/brainsci15030226. PMID 40149748
- See also: Pre-registration of the study — https://osf.io/25afe